CLINICAL TRIAL: NCT00987259
Title: Determination of the Time Course of Myocardial Oedema Post Myocardial Infarction Treated With Primary Angioplasty Using Cardiac Magnetic Resonance Imaging
Brief Title: Myocardial Oedema in Acute Myocardial Infarction (AMI)
Status: Completed | Type: Observational
Sponsor: Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: BLT006964
Record Dates: First submitted 2009-09-29; First posted 2009-09-30 (Estimated); Last update posted 2013-02-01 (Estimated); Status verified 2009-09

CONDITIONS: Myocardial Infarction
Keywords: Myocardial infarction; Myocardial oedema; Magnetic resonance
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Post MI patients: Patients recruited following a successfully reperfused myocardial infarction using primary angioplasty.

SUMMARY:
Despite recent improvements in treatment, myocardial infarction (heart attack) is still a leading cause of illness and death in the UK. Following the acute event, it is difficult to predict which patients are at risk of further problems, such as heart failure and is therefore difficult to know which patients need more aggressive/intensive treatment and monitoring.

There needs to be a test which is safe, reliable and reproducible that can be used shortly after a heart attack to both predict future cardiac events and to allow the efficacy of new treatments to be assessed.

Myocardial oedema (swelling of the heart muscle) has been demonstrated using Cardiac Magnetic Resonance (CMR), to occur following a heart attack and has been suggested as a marker for future cardiac events. The optimum time to perform this scan, the method of data analysis and it's effectiveness as a predictor of future cardiac events has not been adequately assessed.

This trial will assess the amount and natural time-course of oedema in the first 10 days following a heart attack. It will also correlate the amount of oedema with the size of scar (damaged heart muscle) and left ventricular ejection fraction (heart function) at 3 months to assess if it is a predictive marker.

ELIGIBILITY:
Inclusion Criteria:

1. Patients presenting to the London Chest Hospital with acute ST elevation myocardial infarction and treated with primary angioplasty and stent implantation within 12 hours of symptom onset
2. Acute PCI / stent implantation has been successful (residual stenosis visually < 30% and TIMI flow ≥ 2)
3. At the time of inclusion, the patient no longer requires intravenous catecholamines or mechanical hemodynamic support (aortic balloon pump)
4. Serum troponin >1ng/ml 12 hours after onset of pain
5. The patient is able to give written informed consent
6. The patient must be able to understand and communicate in English

Exclusion Criteria:

1. Known cardiomyopathy
2. Previous documented myocardial infarction
3. Previous percutaneous coronary intervention or coronary artery bypass surgery
4. Significant renal dysfunction (EGFR<30)
5. Systemic steroid therapy
6. Current non steroidal anti-inflammatory drug use
7. Chronic inflammatory disease
8. Neoplastic disease without documented remission within the past 5 years
9. Pregnancy
10. Reduced mental capacity leading to inability to obtain informed consent
11. Participation in another clinical trial within the last 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to The London Chest Hospital following an ST elevation myocardial infarction who have been successfully treated with primary angioplasty.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2009-11; Primary Completion 2011-06 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Extent and time course of myocardial oedema over the first 10 days post MI | Days 1, 3 and 10 post MI

SECONDARY OUTCOMES:
Left ventricular ejection fraction and left ventricular scar size at 3 months | 90 days post MI

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R Burchell, BSc, MB BS, Principal Investigator — Bart's and The London NHS Trust, United Kingdom
Locations (1):
- The London Chest Hospital, London, Greater London, United Kingdom

REFERENCES:
- [Background] Higgins CB, Herfkens R, Lipton MJ, Sievers R, Sheldon P, Kaufman L, Crooks LE. Nuclear magnetic resonance imaging of acute myocardial infarction in dogs: alterations in magnetic relaxation times. Am J Cardiol. 1983 Jul;52(1):184-8. doi: 10.1016/0002-9149(83)90093-0. PMID 6858909
- [Background] Laine GA, Granger HJ. Microvascular, interstitial, and lymphatic interactions in normal heart. Am J Physiol. 1985 Oct;249(4 Pt 2):H834-42. doi: 10.1152/ajpheart.1985.249.4.H834. PMID 4051019
- [Background] Nilsson JC, Nielsen G, Groenning BA, Fritz-Hansen T, Sondergaard L, Jensen GB, Larsson HB. Sustained postinfarction myocardial oedema in humans visualised by magnetic resonance imaging. Heart. 2001 Jun;85(6):639-42. doi: 10.1136/heart.85.6.639. PMID 11359743
- [Background] Garcia-Dorado D, Oliveras J, Gili J, Sanz E, Perez-Villa F, Barrabes J, Carreras MJ, Solares J, Soler-Soler J. Analysis of myocardial oedema by magnetic resonance imaging early after coronary artery occlusion with or without reperfusion. Cardiovasc Res. 1993 Aug;27(8):1462-9. doi: 10.1093/cvr/27.8.1462. PMID 8297415
- [Background] Bragadeesh T, Jayaweera AR, Pascotto M, Micari A, Le DE, Kramer CM, Epstein FH, Kaul S. Post-ischaemic myocardial dysfunction (stunning) results from myofibrillar oedema. Heart. 2008 Feb;94(2):166-71. doi: 10.1136/hrt.2006.102434. Epub 2007 Jul 16. PMID 17639092
- [Background] Abdel-Aty H, Boye P, Zagrosek A, Wassmuth R, Kumar A, Messroghli D, Bock P, Dietz R, Friedrich MG, Schulz-Menger J. Diagnostic performance of cardiovascular magnetic resonance in patients with suspected acute myocarditis: comparison of different approaches. J Am Coll Cardiol. 2005 Jun 7;45(11):1815-22. doi: 10.1016/j.jacc.2004.11.069. PMID 15936612
- [Background] Arai AE. Using magnetic resonance imaging to characterize recent myocardial injury: utility in acute coronary syndrome and other clinical scenarios. Circulation. 2008 Aug 19;118(8):795-6. doi: 10.1161/CIRCULATIONAHA.108.797373. No abstract available. PMID 18711021
- [Background] Klem I, Kim RJ. Assessment of microvascular injury after acute myocardial infarction: importance of the area at risk. Nat Clin Pract Cardiovasc Med. 2008 Dec;5(12):756-7. doi: 10.1038/ncpcardio1373. Epub 2008 Oct 14. PMID 18852712
- [Background] Tilak GS, Hsu LY, Hoyt RF Jr, Arai AE, Aletras AH. In vivo T2-weighted magnetic resonance imaging can accurately determine the ischemic area at risk for 2-day-old nonreperfused myocardial infarction. Invest Radiol. 2008 Jan;43(1):7-15. doi: 10.1097/RLI.0b013e3181558822. PMID 18097272
- [Background] Aletras AH, Tilak GS, Natanzon A, Hsu LY, Gonzalez FM, Hoyt RF Jr, Arai AE. Retrospective determination of the area at risk for reperfused acute myocardial infarction with T2-weighted cardiac magnetic resonance imaging: histopathological and displacement encoding with stimulated echoes (DENSE) functional validations. Circulation. 2006 Apr 18;113(15):1865-70. doi: 10.1161/CIRCULATIONAHA.105.576025. Epub 2006 Apr 10. PMID 16606793
- [Background] Friedrich MG, Abdel-Aty H, Taylor A, Schulz-Menger J, Messroghli D, Dietz R. The salvaged area at risk in reperfused acute myocardial infarction as visualized by cardiovascular magnetic resonance. J Am Coll Cardiol. 2008 Apr 22;51(16):1581-7. doi: 10.1016/j.jacc.2008.01.019. PMID 18420102
- [Background] Schulz-Menger J, Gross M, Messroghli D, Uhlich F, Dietz R, Friedrich MG. Cardiovascular magnetic resonance of acute myocardial infarction at a very early stage. J Am Coll Cardiol. 2003 Aug 6;42(3):513-8. doi: 10.1016/s0735-1097(03)00717-4. PMID 12906982
- [Background] Ripa RS, Nilsson JC, Wang Y, Sondergaard L, Jorgensen E, Kastrup J. Short- and long-term changes in myocardial function, morphology, edema, and infarct mass after ST-segment elevation myocardial infarction evaluated by serial magnetic resonance imaging. Am Heart J. 2007 Nov;154(5):929-36. doi: 10.1016/j.ahj.2007.06.038. PMID 17967600